CLINICAL TRIAL: NCT02135146
Title: Evaluating Fluid Strategies in Thoracic Surgery Patients Utilizing a Goal Directed Approach
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-1900; 13-1900 (Other: COMIRB)
Record Dates: First submitted 2014-05-06; First posted 2014-05-09 (Estimated); Results first posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Hypotension; Kidney Injury
Keywords: Hypotension; Kidney injury
MeSH Terms: conditions — Hypotension | interventions — Plasmalyte A; Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plasmalyte 3ml/kg/hr group (Active Comparator)
  Interventions: Drug: Plasmalyte 3ml/kg/hr group
- Plasmalyte 6ml/kg/hr group (Active Comparator)
  Interventions: Drug: Plasmalyte 6ml/kg/hr group

INTERVENTIONS:
Drug: Plasmalyte 3ml/kg/hr group — This group will have intravenous plasmalyte fluid limited to a rate of 3 ml/kg/hr. and a nexfin monitor placed on them
  Arms: Plasmalyte 3ml/kg/hr group
Drug: Plasmalyte 6ml/kg/hr group — This group will have intravenous plasmalyte fluid limited to a rate of 6 ml/kg/hr. and a Nexfix Monitor placed on them
  Arms: Plasmalyte 6ml/kg/hr group

SUMMARY:
The purpose of this study is to conduct a prospective, randomized, controlled trial comparing a restrictive vs. conservative fluid strategy in thoracic surgery patients. Excessive perioperative fluid has been retrospectively implicated in the development postoperative acute lung injury (PALI) and pulmonary edema following lung resection. However, fluid restriction in these patients is not without risk and may compromise end organ perfusion (i.e. acute kidney injury). The hypothesis is that a conservative fluid approach in thoracic surgery patients will result in better end organ perfusion with fewer occasions of acute kidney injury (AKI) without causing an increase in postoperative acute lung injury or pulmonary edema.

ELIGIBILITY:
Inclusion Criteria:

* between 18-89 years of age
* undergoing pulmonary lobectomy with open or video assisted thoracotomy

Exclusion Criteria:

* patient refusal
* pregnancy
* cardiac arrhythmia
* pacemaker dependency
* severe aortic insufficiency
* idiopathic hypertrophic subaortic stenosis
* prisoners
* decisionally challenged
* patients that refuse to receive intravenous fluid products made from human plasma (Albumin 5%)
* patients with skin infection or breakdown on their fingers
* severe peripheral vascular disease
* evidence of compromised finger perfusion will be excluded

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamas Seres, M.D., PH.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Plasmalyte 3ml/kg/hr Group | Plasmalyte 6ml/kg/hr Group
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Plasmalyte 3ml/kg/hr Group | Plasmalyte 6ml/kg/hr Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (9.2) | 65.1 (12.1) | 63.6 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 4 | 1 | 5
ASA Score [Count of Participants; unit: Participants] — The American Society of Anesthesiology (ASA) Physical Status Classification of the patient's present physical condition on a scale from 1-6 classifications are as follows: ASA 1. Normal healthy patient.
  ASA 2. Patient with mild systemic disease. ASA 3. Patient with severe systemic disease. ASA 4. Patient with severe systemic disease that is a constant threat to life. ASA 5. Moribund patient who is not expected to survive without the operation. ASA 6. Declared brain-dead patient whose organs are being removed for donor purposes.
  Participants
    ASA 2 | 9 | 5 | 14
    ASA 3 | 11 | 15 | 26
Body Weight [Mean (Standard Deviation); unit: kg] | 58.8 (10.9) | 65.2 (12.1) | 62.02 (11.9)
Ideal Body Weight [Mean (Standard Deviation); unit: kg] | 57.9 (8.5) | 57.16 (5.5) | 57.5 (7.1)
Height [Mean (Standard Deviation); unit: cm] | 165.1 (7.9) | 165 (5.9) | 165.05 (6.8)
BMI [Mean (Standard Deviation); unit: kg/m2] — Body Mass Index (BMI) is weight in kilograms divided by the square of height in meters. Scores between 18.5 and 24.9 indicate healthy body weights. Higher scores indicate higher body weights.
  kg/m2 | 21.5 (3.2) | 24.1 (4.9) | 22.8 (4.3)
Epidural [Count of Participants; unit: Participants] | 4 | 3 | 7
Smoker [Count of Participants; unit: Participants] | 9 | 9 | 18
Chronic Obstructive Pulmonary Disease (COPD) [Count of Participants; unit: Participants] | 5 | 0 | 5
Asthma [Count of Participants; unit: Participants] | 3 | 2 | 5
Pulmonary Hypertension [Count of Participants; unit: Participants] | 0 | 0 | 0
Coronary Artery Disease (CAD) [Count of Participants; unit: Participants] | 1 | 1 | 2
Hypertension (HTN) [Count of Participants; unit: Participants] | 6 | 4 | 10
Heart Disease [Count of Participants; unit: Participants] | 0 | 1 | 1
Peripheral Vascular Disease (PVD) [Count of Participants; unit: Participants] | 0 | 0 | 0
Diabetes [Count of Participants; unit: Participants] | 3 | 0 | 3
Hepatitis [Count of Participants; unit: Participants] | 3 | 0 | 3
Chronic Kidney Disease (CKD) [Count of Participants; unit: Participants] | 0 | 0 | 0
Seizure [Count of Participants; unit: Participants] | 1 | 0 | 1
Lung Cancer [Count of Participants; unit: Participants] | 5 | 7 | 12
Chronic Lung Infection [Count of Participants; unit: Participants] | 15 | 13 | 28
Surgical Procedure (Video-Assisted Thoracoscopic Surgery-VATS) [Count of Participants; unit: Participants] | 18 | 19 | 37
Procedure Duration [Mean (Standard Deviation); unit: min] | 162.1 (75.1) | 153.4 (62.7) | 157.8 (68.5)
Anesthesia Duration [Mean (Standard Deviation); unit: min] | 206.6 (79.4) | 198.9 (67.4) | 202.7 (72.8)
Creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.86 (0.22) | 0.84 (0.17) | 0.85 (0.195)

OUTCOME MEASURES:

1. Primary Outcome: Development of Renal Injury
Description: Acute renal injury as defined by the American Kidney Injury Network (AKIN) criteria in the first 72 hours postoperatively (serum creatinine levels). The AKIN scale will be used to assess the presence and severity of acute kidney injury (AKI). The AKIN is a classification/staging system of acute kidney injury developed by the Acute Kidney Injury Network which uses changes in serum creatinine (SCr) and urine output to assess AKI. Stages of acute kidney injury are defined as 1, 2, or 3, with 3 indicating the most severe AKI.
  (1) Increase ≥ 0.3 mg per dL (26.52 μmol per L) or ≥ 1.5- to twofold from baseline. (2) Increase > two- to threefold from baseline. (3) Increase > threefold from baseline or ≥ 4.0 mg per dL (353.60 μmol per L) with an acute rise of at least 0.5 mg per dL (44.20 μmol per L).
Time Frame: Post-op up to 72 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Plasmalyte 3ml/kg/hr Group | Plasmalyte 6ml/kg/hr Group
Number analyzed (Participants) | 20 | 20
mg/dL | 0.8 (0.25) | 0.74 (0.14)
Statistical Analysis 1: Comparison: Plasmalyte 3ml/kg/hr Group; Test type: Superiority; p = 0.31, t-test, 2 sided
Statistical Analysis 2: Comparison: Plasmalyte 6ml/kg/hr Group; Test type: Superiority; p = 0.07, t-test, 2 sided

2. Primary Outcome: Development of Pulmonary Edema
Description: The number of participants diagnosed with mild to severe pulmonary edema at any time up to 72 hours after surgery is reported.
Time Frame: Post-op up to 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Plasmalyte 3ml/kg/hr Group | Plasmalyte 6ml/kg/hr Group
Number analyzed (Participants) | 20 | 20
Participants | 4 | 3

3. Secondary Outcome: Length of Surgical Intensive Unit Stay/Hospital Stay
Description: Length of Surgical Intensive Unit Stay/Hospital Stay
Time Frame: Up to 7 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Plasmalyte 3ml/kg/hr Group | Plasmalyte 6ml/kg/hr Group
Number analyzed (Participants) | 20 | 20
days | 0.6 (1.5) | 0.2 (0.7)

4. Secondary Outcome: Removal of Chest Tubes
Description: Time to removal of Chest Tubes
Time Frame: Post-op up to 48 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Plasmalyte 3ml/kg/hr Group | Plasmalyte 6ml/kg/hr Group
Number analyzed (Participants) | 20 | 20
minutes | 3.5 (2.5) | 3.7 (3.9)

5. Secondary Outcome: Development of Morbidity
Description: Development of Morbidity, including: acute lung injury, Acute Respiratory Distress, Deep Vein Thrombus, infection, delirium
Time Frame: Up to 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Plasmalyte 3ml/kg/hr Group | Plasmalyte 6ml/kg/hr Group
Number analyzed (Participants) | 20 | 20
Participants | 4 | 5

6. Secondary Outcome: Death
Description: Death
Time Frame: Assessed up to 30 days Post-op
Population: Missing participants lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Plasmalyte 3ml/kg/hr Group | Plasmalyte 6ml/kg/hr Group
Number analyzed (Participants) | 9 | 11
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Plasmalyte 3ml/kg/hr Group | Plasmalyte 6ml/kg/hr Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 4/20 | 5/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plasmalyte 3ml/kg/hr Group (N=20) | Plasmalyte 6ml/kg/hr Group (N=20)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (SVT) (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes